CLINICAL TRIAL: NCT01862224
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Synovial Biopsy Study of JNJ-38518168 in Subjects With Active Rheumatoid Arthritis Despite Methotrexate Therapy
Brief Title: A Synovial Biopsy Study of JNJ-38518168 in Participants With Active Rheumatoid Arthritis Despite Methotrexate Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was stopped due to lack of efficacy in a study conducted in a similar population,38518168ARA2002-NCT01679951.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR100963; 38518168ARA2003 (Other: Janssen Research & Development, LLC); 2011-006325-18 (EudraCT Number)
Record Dates: First submitted 2013-05-02; First posted 2013-05-24 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Active rheumatoid arthritis despite methotrexate therapy; JNJ-38518168; Synovial
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- JNJ-38518168 (Experimental): JNJ-38518168 30 mg once daily for 52 weeks.
  Interventions: Drug: JNJ-38518168; Drug: Methotrexate
- Placebo/JNJ-38518168 (Placebo Comparator): Matching placebo once daily for 12 weeks followed by JNJ-38518168 30 mg once daily for 40 weeks.
  Interventions: Drug: JNJ-38518168; Drug: Placebo; Drug: Methotrexate

INTERVENTIONS:
Drug: JNJ-38518168 — JNJ-38518168 30 mg once daily, Week 0 to Week 52.
Drug: Placebo — Matching placebo once daily (Week 0 to Week 12).
  Arms: Placebo/JNJ-38518168
Drug: Methotrexate — All participants will continue receiving methotrexate up to Week 12. After Week 12, the dose of methotrexate may be adjusted as per Investigator's discretion.

SUMMARY:
The purpose of this study is to assess the impact of JNJ-38518168 on rheumatoid arthritis (RA) disease-related biomarkers in synovial biopsy tissue and blood in participants with active RA despite methotrexate (MTX) therapy and to assess the safety and tolerability of JNJ-38518168 over one year.

DETAILED DESCRIPTION:
This is a randomized (participants assigned to treatment by chance), double-blind (participants and study personnel will not know what treatment is being given), placebo-controlled (a placebo appears identical to a study drug, but contains no active ingredients), parallel-group (treatments will be given to groups of participants at the same time) study. Participants will be randomly assigned in a 3:1 ratio to receive either JNJ-38518168 for 52 weeks or receive matching placebo for 12 weeks, followed by JNJ-38518168 for 40 weeks. The total duration of participation will be approximately 60 weeks for all participants, including a screening visit and follow-up visits. Safety and tolerability of JNJ-38518168 will be evaluated by monitoring adverse events reported by participants throughout the study . In addition, results from clinical laboratory tests, electrocardiograms, vital signs measurements, and physical examinations performed during the study will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Have had rheumatoid arthritis (RA) for at least 6 months prior to the date of signing the informed consent at screening
* Be positive for either anti-cyclic citrullinated peptide (anti-CCP) antibody or rheumatoid factor (RF) in serum at screening
* Have active RA defined for the purpose of this study as persistent disease activity with both of the following criteria: At least 4 swollen and 4 tender joints using a 66/68 joint count. At the time of screening, one of the tender or swollen joints or both must include the non-prosthetic knee to be biopsied; and serum C-reactive protein (CRP_ ≥ 0.60 mg/dL at screening
* Have been treated with and tolerated oral methotrexate (MTX) treatment at doses from 10 mg/week to 25 mg/week inclusive, for a minimum of 3 months prior to the date of signing the informed consent at screening and must have a stable MTX dose for a minimum of 8 weeks prior to the date of signing the informed consent at screening and continue to receive the same MTX dose at Week 0
* If using nonsteroidal anti-inflammatory drugs (NSAIDs) or other analgesics (pain relievers) regularly for RA, the participant must have been on a stable dose for at least 2 weeks prior to the first administration of study agent. If not using NSAIDs or other analgesics for RA at Week 0, the participant must have not received NSAIDs or other analgesics for RA for at least 2 weeks prior to the first administration of study agent

Exclusion Criteria:

* Has inflammatory diseases other than RA
* Has a history of juvenile idiopathic arthritis (JIA)
* Has current signs or symptoms of liver or renal insufficiency or cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, psychiatric, or metabolic disturbances that are severe, progressive, or uncontrolled

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Assessment of rheumatoid arthritis (RA) biomarkers | Up to Week 52
  Biomarkers may include, but are not limited to, inflammatory markers and cytokines; synovium/cartilage/bone markers; and gene expression profiles.

SECONDARY OUTCOMES:
Number of participants reporting adverse events as a measure of safety and tolerability | Up to Week 56

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (2):
- Frederick, Maryland, United States
- Chisinau, Moldova